CLINICAL TRIAL: NCT00574821
Title: Assessing the Utility of Magnetocardiography in Patients With Hypertrophic Cardiomyopathy
Brief Title: Use of Magnetic Field Mapping in the Evaluation of Patients With Hypertrophic Heart Disease (Thick Heart Muscle)
Status: Withdrawn | Type: Observational
Why Stopped: sponsor funding
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: CardioMag Imaging (Industry)
Responsible Party: Kirsten Tolstrup, MD, Cedars-Sinai Medical Center
Other Study IDs: 11958
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic Cardiomyopathy(HCM); Magnetocardiography (MCG)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to further establish the diagnostic use of magnetocardiography (MCG) in patients with hypertrophic cardiomyopathy (HCM). The use of MCG has not been extensively studied in these patients. This pilot study will serve to further characterize abnormalities found on MCG in comparison to patients without hypertrophic cardiomyopathy. Additionally, the study will be used to understand whether MCG has any additional diagnostic utility in offering clinicians insight on the patient's disease state, thereby aiding in the development of treatment plans.

This research study is designed to test the effectiveness of the investigational use of magnetocardiography in patients with hypertrophic cardiomyopathy. The device itself has been approved by the U.S Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Patients with hypertrophic cardiomyopathy (HCM) have a gene mutation that results in excessive thickening of heart muscle. Due to this abnormality these patients often present with voltage changes on electrocardiograms (ECG) suggestive of abnormal electrical conduction. The use of magnetocardiography (MCG) in these patients has yet to be extensively studied. Magnetocardiography (MCG) is a safe, non-invasive, and FDA approved technology that can be used to detect weak magnetic fields generated by the heart. The goal of this pilot study is to determine common MCG findings in patients with HCM, while establishing the role that MCG has in the evaluation and treatment of these patients.

We will enroll a total of twenty patients identified to have hypertrophic cardiomyopathy by cardiologists at our facility. As patients' enroll in the study, data will be collected prospectively. We will continue to follow up on patients over the course of 1 year from the date of their initial enrollment. Once a patient has been identified as a candidate for this study, they will be instructed about the risks and benefits of undergoing participation. Informed consent to participate in the study will be obtained for each patient.

We will obtain basic demographic information on our patients including sex, age, race, weight, height, and other co-morbidities and cardiovascular risk factors including, but not limited to family history of syncope, sudden cardiac death, chest pain, or shortness of breath. Information in regards to symptoms experienced, onset of symptoms, previous and current diagnostic workup included blood work and cardiac scans, and current/past treatments will also be recorded. A list of medications will be recorded.

Prior to the MCG scan, the patient will be instructed to wear only non-metallic containing clothing. Patients's will then be requested to lie still on a table for a duration of 6 minutes, while undergoing a magnetocardiography scan. In addition to the MCG, the patient's blood pressure and a 12-lead electrocardiogram will be obtained. Most patients will also have a complete 2D echocardiogram which will require the patient to lie down on a table while an ultrasound probe is placed on the left side of the chest resulting in an image of the heart on a computer screen. In addition to the above, if clinically indicated patients may have blood draws taken at the discretion of their cardiologist. These blood draws may be used to obtain lipid levels, cardiac biomarkers, and natriuretic peptide assays (used to evaluate heart failure).

Once a patient has completed an initial assessment and scan, we will ask the patient to return for follow up visits at 3 months and 1 year for repeat MCG. A 2D ECHO will be obtained at 3 months if clinically indicated, and at 1 year. In addition, we are asking for follow up scans if the patient presents with any cardiac symptoms such as chest pain, shortness of breath, or fainting Follow up phone interview will occur at 6 months. We will ask information regarding symptoms, treatments, hospital admissions, cardiologist visits, and any subsequent diagnostic testing performed including ECGs, transthoracic echos, transesophageal echos, exercise/chemical stress testing, angiograms, and cardiac catheterizations.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient that is hemodynamically stable and is identified to have hypertrophic cardiomyopathy based on prior symptoms, 2D ECHO findings, genetic testing, and/or ECG voltage criteria.
2. Patients that have signed informed consent after understanding the risks and benefits of participation. Individual age 16-17 with the consent and approval of a parent and /or legal guardian.

Exclusion Criteria:

1. Patients with prior history of myocardial infarction, CAD demonstrated by stress test or angiogram, and/or CABG will be excluded from this study.
2. Any patient that has undergone invasive treatment at the time of enrollment including procedures such as myomectomy and/or septal ablation. However, already enrolled subjects who have these procedures post-enrollment into the study will be eligible for future scans.
3. Patients encountering any significant symptoms, chest pain, or who are hemodynamically unstable.
4. Any patient with an ICD or pacemaker.
5. Patients who are underage and do not have the consent of a parent and/or legal guardian.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will enroll a total of twenty patients identified to have hypertrophic cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tolstrup, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States